CLINICAL TRIAL: NCT03803631
Title: CNV in AMD Analyzed by OCT Angiography Under IntravitreaL Eylea (COCTAEyl)
Acronym: COCTAEyl
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: COCTAEyl
Record Dates: First submitted 2018-09-11; First posted 2019-01-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: AMD; Exudative Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to analyze a new noninvasive imaging examination, OCT angiography, in the evaluation of neovascular remodeling and early signs of recurrence of wet AMD undergoing treatment on OCTA and to correlate OCTA findings with SD-OCT findings.

ELIGIBILITY:
Inclusion Criteria:

* Naïve patients
* Type 1 or type 2 Choroidal NeoVascularization (CNV)
* Age ≥ 55 years
* Presence of subfoveal CNV secondary to Age-related Macular Degeneration (AMD)
* At the time of inclusion, multimodal imaging should reveal exudative features
* Exudative AMD diagnosis established between 1 and 7 days before inclusion
* Monitored monthly
* Loading phase then bimonthly retreatment.
* Signed Informed Consent.
* Patient covered by the French Health Insurance

Exclusion Criteria:

* Polypoidal choroidal vasculopathy
* Type 3 neovascularization
* Choroidal neovascularization attributable to causes other than AMD
* Macular hematoma
* Pigment epithelial detachment higher than 150µm
* Fibrosis > 50% lesion on fundus color photography, fibroglial scar
* Media opacity annoying acquisition
* Retinal vascular occlusion
* Diabetic retinopathy
* Adult-onset foveomacular vitelliform dystrophy and other pattern dystrophies,
* Refractive error >-6D
* Active intraocular inflammation in the study eye
* Patient who does not meet the local indication criteria for Eylea® treatment. Contraindications listed in the SmPCs must be taken into account
* Patient taking part in an interventional study at the time of enrolment.
* Any history of allergy to the antiseptic used during preparation of the eye for the IVT injection in the investigational site (e.g. povidone iodine or chlorhexidine).
* Pregnant and lactating women
* Stroke and/or myocardial infarction 3 months before inclusion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wet-AMD (NVC type 1 or 2) diagnosed maximum one week before inclusion and for whom Aflibercept in intra-vitreal injection technic has been prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
presence of flow on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 13
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time

SECONDARY OUTCOMES:
presence of flow on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of collaterals on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of peripheral arcade on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of arteriolization on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of vascular loops on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of dark halo on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of feeder vessel on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
presence of flow void on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular area on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | baseline
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 1
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 2
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 3
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 4
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 5
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 6
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 7
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 8
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 9
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 10
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 11
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
measure of neovascular density on OCTA | at month 12
  high flow on OCTA corresponding to the neovascular network with vascular remodeling over time
Intraretinal and/or subretinal fluid in SD-OCT | at month 13
Intraretinal and/or subretinal fluid in SD-OCT | at baseline
Intraretinal and/or subretinal fluid in SD-OCT | at month 1
Intraretinal and/or subretinal fluid in SD-OCT | at month 2
Intraretinal and/or subretinal fluid in SD-OCT | at month 3
Intraretinal and/or subretinal fluid in SD-OCT | at month 4
Intraretinal and/or subretinal fluid in SD-OCT | at month 5
Intraretinal and/or subretinal fluid in SD-OCT | at month 6
Intraretinal and/or subretinal fluid in SD-OCT | at month 7
Intraretinal and/or subretinal fluid in SD-OCT | at month 8
Intraretinal and/or subretinal fluid in SD-OCT | at month 9
Intraretinal and/or subretinal fluid in SD-OCT | at month 10
Intraretinal and/or subretinal fluid in SD-OCT | at month 11
Intraretinal and/or subretinal fluid in SD-OCT | at month 12
visual acuity in logmar | at baseline
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 1
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 2
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 3
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 4
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 5
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 6
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 7
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 8
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 9
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 10
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 11
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 12
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
visual acuity in logmar | at month 13
  Measure of best-corrected visual acuity (BCVA) measured on ETDRS
presence or abscence of hemorrhage, fibrosis and atrophy on fundus color photography | at 1 months
presence or abscence of hemorrhage on fundus color photography | at 1 months
presence or abscence of fibrosis on fundus color photography | at 1 months
presence or abscence of atrophy on fundus color photography | at 1 months
presence or abscence of hemorrhage on fundus color photography | at 13 months
presence or abscence of fibrosis on fundus color photography | at 13 months
presence or abscence of atrophy on fundus color photography | at 13 months
type of choroidal neovascularization on fluorescein angiography (type 1, type 2 or mixed lesions) | Baseline
type of choroidal neovascularization on fluorescein angiography (type 1, type 2 or mixed lesions) | at month 13
type of choroidal neovascularization on indocyanine green angiography (type 1, type 2 or mixed lesions) | baseline
type of choroidal neovascularization on indocyanine green angiography (type 1, type 2 or mixed lesions) | at month 13
choroidal thickness on EDI-OCT | monthly during 13 months
type of choroidal neovascularization on SD-OCT (type 1, type 2 or mixed lesions) | monthly during 13 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Pellegrin, CHU de Bordeaux, Bordeaux
  - CHI de Créteil, Créteil
  - Hôpital La Croix Rousse, Lyon
  - Hôpital Lariboisière, APHP, Paris
  - Centre Ophtalmologique d'Imagerie et de Laser,, Paris

IPD SHARING:
Plan to Share IPD: Undecided